CLINICAL TRIAL: NCT00492310
Title: Yoga for Women Attempting Smoking Cessation: an Initial Investigation
Brief Title: Yoga for Women Attempting Smoking Cessation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Beth Bock, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT003669-01 (NIH); R21AT003669-01 (NIH)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Smoking
Keywords: Smoking; tobacco; women; yoga
MeSH Terms: conditions — Smoking | interventions — Yoga; Cognitive Behavioral Therapy; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive-behavioral smoking cessation with yoga
  Interventions: Behavioral: yoga; Behavioral: cognitive therapy
- 2 (Active Comparator): smoking cessation with twice weekly wellness program
  Interventions: Behavioral: cognitive therapy; Behavioral: wellness

INTERVENTIONS:
Behavioral: yoga — vinyasa yoga
  Arms: 1
Behavioral: cognitive therapy — cognitive behavioral therapy once weekly
Behavioral: yoga — vinyasa yoga twice weekly with smoking cessation once weekly
  Arms: 1
Behavioral: wellness — wellness program with smoking cessation
  Arms: 2

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability and initial effectiveness of adding yoga to a traditional, group-based treatment for smoking cessation for women smokers.

DETAILED DESCRIPTION:
Smoking is the leading preventable cause of morbidity and mortality among women in the US. Quitting smoking may be especially problematic for women. As a form of exercise, yoga shares many of the same properties as traditional (Western) aerobic exercise which our previous research has shown to be an effective addition to smoking cessation. Yoga may also offer other benefits that may make it an especially effective complimentary treatment for women who are attempting to quit smoking.

In this study we will recruit two cohorts of 30 women smokers and provide cognitive-behavioral therapy for smoking cessation once weekly for 12 weeks. In addition, participants will be randomly assigned them to receive either; (1) Yoga or (2) a Wellness program (contact-control), twice weekly during the program. All participants will be assessed for changes in smoking behavior, psychosocial variables relevant to smoking cessation and other psychological constructs that may act as mechanisms of action (mediators) of yoga and smoking cessation. These variables include; weight concerns, perceived stress, mindfulness, self-esteem, quality of life and group cohesion. Interviews will be used to collect qualitative data at the end of each cohort. The proposed study is designed to provide information necessary to establish several research fundamentals necessary to support a full scale efficacy trial. These include: 1) establishing intervention feasibility and acceptability in the target population, 2) piloting recruitment and retention procedures and identifying barriers to participation, 3) obtaining qualitative feedback from participants to enhance treatment content and/or design, 4) establishing anticipated effect size estimates, and 5) identifying likely mechanisms of action that may be responsible for intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

Female, Age 18-65, Cigarette smoking 10 or more per day for more than 1 year, sedentary (not exercising more than 2 days per week)

Exclusion Criteria:

Major depression, Hypertension, Current yoga practice, Current mind/body therapies

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
smoking cessation: 7-day point prevalence abstinence | 6 months

SECONDARY OUTCOMES:
Acceptability: recruitment, retention, adherence to protocol | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Beth C Bock, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Bock BC, Morrow KM, Becker BM, Williams DM, Tremont G, Gaskins RB, Jennings E, Fava J, Marcus BH. Yoga as a complementary treatment for smoking cessation: rationale, study design and participant characteristics of the Quitting-in-Balance study. BMC Complement Altern Med. 2010 Apr 29;10:14. doi: 10.1186/1472-6882-10-14. PMID 20429895